CLINICAL TRIAL: NCT00341861
Title: Interdisciplinary Case-Control Study of Bladder Cancer in Spain
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999038; OH99-C-N038
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Occupational and Environmental Risks; Lifestyle Factors; Epidemiology; Genetic Susceptibility
MeSH Terms: conditions — Urinary Bladder Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The incidence rate of bladder cancer in the Barcelona area of Spain is almost identical to that of the U.S. Cigarette smoking has been identified as the most significant risk factor for bladder cancer, followed by occupational exposures to chemicals such as aromatic amines and their derivatives, diesel exhaust, oil mist, pesticides, and polynuclear aromatic hydrocarbons. A variety of non-occupational exposures have been suggested as potential risk factors as well, including smoking black vs. blond tobacco, dietary factors, certain medications and medical conditions, chlorination by-products in drinking water, and fluid intake. Various genetic polymorphisms also appear to affect bladder cancer risk. Research is needed to further explore hypotheses generated by previous etiologic studies of bladder cancer. An on-going study of bladder cancer survival by the Institut Municipal d'Investigacio Medica in Spain provides an excellent opportunity for NCI to perform such research. NCI will build upon the ongoing study by funding an interdisciplinary case-control component to evaluate bladder cancer risk in relation to various external factors (e.g., occupational and environmental exposure) and host factors (e.g., genetic susceptibility markers, and early effect markers). This hospital-based case-control study will involve personal interviews using a state-of-the-art, computer assisted technique, and collection of blood and toenail samples from participants.

DETAILED DESCRIPTION:
The incidence rate of bladder cancer in the Barcelona area of Spain is almost identical to that of the U.S. Cigarette smoking has been identified as the most significant risk factor for bladder cancer, followed by occupational exposures to chemicals such as aromatic amines and their derivatives, diesel exhaust, oil mist, pesticides, and polynuclear aromatic hydrocarbons. A variety of non-occupational exposures have been suggested as potential risk factors as well, including smoking black vs. blond tobacco, dietary factors, certain medications and medical conditions, chlorination by-products in drinking water, and fluid intake. Various genetic polymorphisms also appear to affect bladder cancer risk. Research is needed to further explore hypotheses generated by previous etiologic studies of bladder cancer. An ongoing study of bladder cancer survival by the Institut Municipal d'Investigacio Medica in Spain provides an excellent opportunity for NCI to perform such research. NCI will build upon the ongoing study by funding an interdisciplinary case-control component to evaluate bladder cancer risk in relation to various external factors (e.g., occupational and environmental exposure) and host factors (e.g., genetic susceptibility marker, and early effect markers). This hospital-based case-control study will involve personal interviews using a state-of-the-art, computer-assisted technique, and collection of blood and toenail samples from participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

All histologically confirmed cases of carcinoma of the bladder including carcinoma in situ at the 21 centers.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a hospital-based case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 2925 (Actual)
Dates: Start 1998-09-01 (Actual); Primary Completion 2012-12-04 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Bladder Cancer | 1998-2000
  Incident bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Debra Silverman, D.Sc., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Institut Municipal d'Investigacio Medica, Barcelona, Spain

REFERENCES:
- [Background] Agundez JA, Martinez C, Olivera M, Ledesma MC, Ladero JM, Benitez J. Molecular analysis of the arylamine N-acetyltransferase polymorphism in a Spanish population. Clin Pharmacol Ther. 1994 Aug;56(2):202-9. doi: 10.1038/clpt.1994.124. PMID 8062497
- [Background] Babu SR, Lakshmi VM, Huang GP, Zenser TV, Davis BB. Glucuronide conjugates of 4-aminobiphenyl and its N-hydroxy metabolites. pH stability and synthesis by human and dog liver. Biochem Pharmacol. 1996 Jun 28;51(12):1679-85. doi: 10.1016/0006-2952(96)00165-7. PMID 8687483
- [Background] Badawi AF, Hirvonen A, Bell DA, Lang NP, Kadlubar FF. Role of aromatic amine acetyltransferases, NAT1 and NAT2, in carcinogen-DNA adduct formation in the human urinary bladder. Cancer Res. 1995 Nov 15;55(22):5230-7. PMID 7585581